CLINICAL TRIAL: NCT01205152
Title: Extension Study of ENB-0040 (Human Recombinant Tissue-Nonspecific Alkaline Phosphatase Fusion Protein) in Severely Affected Infants and Young Children With Hypophosphatasia (HPP)
Brief Title: Extension Study of Protocol ENB-002-08 - Study of Asfotase Alfa in Infants and Young Children With Hypophosphatasia (HPP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENB-003-08; FD-R-003745-03 (Other Grant/Funding Number: Office of Orphan Product Development)
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Hypophosphatasia
Keywords: Hypophosphatasia; HPP; Bone disease; Soft bones; Low alkaline phosphatase; Genetic metabolic disorder; Alkaline phosphatase; Tissue non-specific alkaline phosphatase; Rickets; Osteomalacia
MeSH Terms: conditions — Hypophosphatasia; Bone Diseases; Rickets; Osteomalacia | interventions — asfotase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- asfotase alfa (Experimental): An initial single intravenous (IV) infusion of 2 mg/kg asfotase alfa, followed by subcutaneous (SC) injections of 1 mg/kg asfotase alfa 3 times per week
  Interventions: Biological: asfotase alfa

INTERVENTIONS:
Biological: asfotase alfa
  Other Names: ENB-0040

SUMMARY:
This clinical trial studied the long term safety and efficacy of asfotase alfa in infants and young children with infantile onset HPP who completed study ENB-002-08 (NCT00744042).

Partial funding for this study was provided by the Office of Orphan Product Development (OOPD).

DETAILED DESCRIPTION:
Asfotase Alfa was formerly referred to as ENB-0040

Hypophosphatasia (HPP) is a life-threatening, genetic, and ultra-rare metabolic disease characterized by defective bone mineralization and impaired phosphate and calcium regulation that can lead to progressive damage to multiple vital organs, including destruction and deformity of bones, profound muscle weakness, seizures, impaired renal function, and respiratory failure. There are limited data available on the natural course of this disease over time, particularly in patients with the juvenile-onset form.

ELIGIBILITY:
Inclusion Criteria

* Patient completed participation in ENB-002-08 (NCT00744042)
* Written informed consent by parent or other legal guardian prior to any study procedures being performed
* Parent or other legal guardian willing to comply with study requirements

Exclusion Criteria

* History of sensitivity to any of the constituents of the study drug
* Clinically significant disease that precludes study participation
* Enrollment in any study (other than ENB-002-08) involving an investigational drug, device, or treatment for HPP (e.g., bone marrow transplantation)

Ages: 24 Weeks to 42 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2009-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (5):
  - Alfred I. DuPont Hospital for Children, Wilmington, Delaware
  - St. John's Medical Research Institute, Springfield, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - St. Vincent Hospital, Green Bay, Wisconsin
- Tawam Hospital, Al Ain City, Abu Dhabi Emirate, United Arab Emirates
- United Kingdom (2):
  - Royal Maternity Hospital, Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Sheffield Children's Hospital, Sheffield

REFERENCES:
- [Derived] Padidela R, Yates R, Benscoter D, McPhail G, Chan E, Nichani J, Mughal MZ, Myer C 4th, Narayan O, Nissenbaum C, Wilkinson S, Zhou S, Saal HM. Characterization of tracheobronchomalacia in infants with hypophosphatasia. Orphanet J Rare Dis. 2020 Aug 6;15(1):204. doi: 10.1186/s13023-020-01483-9. PMID 32762706
- [Derived] Whyte MP, Simmons JH, Moseley S, Fujita KP, Bishop N, Salman NJ, Taylor J, Phillips D, McGinn M, McAlister WH. Asfotase alfa for infants and young children with hypophosphatasia: 7 year outcomes of a single-arm, open-label, phase 2 extension trial. Lancet Diabetes Endocrinol. 2019 Feb;7(2):93-105. doi: 10.1016/S2213-8587(18)30307-3. Epub 2018 Dec 14. PMID 30558909
- [Derived] Whyte MP, Rockman-Greenberg C, Ozono K, Riese R, Moseley S, Melian A, Thompson DD, Bishop N, Hofmann C. Asfotase Alfa Treatment Improves Survival for Perinatal and Infantile Hypophosphatasia. J Clin Endocrinol Metab. 2016 Jan;101(1):334-42. doi: 10.1210/jc.2015-3462. Epub 2015 Nov 3. PMID 26529632
- See also: Hypophosphatasia Website — http://www.hypophosphatasia.com
- See also: Hypophosphatasia Website for Healthcare Providers — http://www.hypophosphatasia.com/hcp/
- See also: HPP support group — http://www.magicfoundation.org
- See also: US Hypophosphatasia Group (Soft Bones) — http://www.softbones.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The main criteria for inclusion in Study ENB-002-08 were male and female patients </= 36 months of age, with severe infantile-onset HPP (symptom onset before 6 months of age) who were medically stable (ventilator support was allowed). To enter extension Study ENB-003-08, parent/guardian had to consent and patient had to complete Study ENB-002-08.
Period: Overall Study
Arm/Group | Asfotase Alfa
Started | 10
Completed | 9
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Of the 11 patients who were enrolled in Study ENB-002-08, 10 patients completed Study ENB-002-08 and were enrolled in extension study ENB-003-08.
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Mean (SD) age at time of first dose in ENB-002-08 (NCT00744042)
  weeks | 56.44 (61.888)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Long-term Tolerability of Subcutaneous (SC) Asfotase Alfa
Description: Outcome measure is the number of patients with 1 or more treatment-emergent adverse event. The time period is from Baseline in the ENB-003-08 study to the end of the ENB-003-08 study.
Time Frame: 84 months
Population: Full Analysis Set (All 10 patients enrolled in Study ENB-003-08)
Measure: Count of Participants; unit: Participants
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 10
Participants | 10

2. Primary Outcome: Long-term Efficacy of Asfotase Alfa in Treating Rickets in Infants and Young Children With Hypophosphatasia (HPP).
Description: Outcome measure is the evaluation of radiographic change in rickets severity using a qualitative Radiographic Global Impression of Change (RGI-C) Scale. Skeletal radiographs obtained at the patient's last assessment were compared with skeletal radiographs obtained before initiation of treatment (Baseline in Study ENB-002-08 [NCT00744042]). The RGI-C is a 7-point rating scale that ranges from -3 (indicative of severe worsening of HPP-associated rickets) to +3 (indicative of complete or near complete healing of HPP-associated rickets).
  The time period is pre-dose (Baseline from ENB-002-08 study) to the last assessment for each patient in the ENB-003-08 study, which represents up to 90 months of exposure for the combined studies.
Time Frame: Up to 90 Months
Population: Full Analysis Set (All 10 patients enrolled in Study ENB-003-08)
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 10
scores on a scale | 2.00 [2.00 to 3.00]
Statistical Analysis 1: Comparison: Asfotase Alfa; Change is relative to Baseline in Study ENB-002-08 (NCT00744042). The RGI-C score represents evaluation of skeletal X-rays at each post-treatment study timepoint compared with pre-treatment X-rays from Study ENB-002-08 using an ordinal scale. Therefore, an RGI-C score is not applicable for radiographs obtained at Baseline; Test type: Other; p = 0.0020, Wilcoxon signed-rank test — Two-sided with p-value threshold <0.05 for statistical significance

3. Secondary Outcome: Long-term Pharmacodynamics (PD) of SC Asfotase Alfa: Plasma Inorganic Pyrophosphate (PPi) Levels
Description: Outcome measure is the change from Baseline in plasma inorganic pyrophosphate (PPi) levels. The time period is pre-dose (Baseline from the ENB-002-08 study [NCT00744042]) to the last assessment for each patient in the ENB-003-08 study, which represents up to 90 months of exposure for the combined studies.
Time Frame: Up to 90 Months
Population: Full Analysis Set (All 10 patients enrolled in Study ENB-003-08). Change from Baseline could not be calculated for 3 patients due to non-evaluable samples at Baseline.
Measure: Median (Full Range); unit: uM
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 7
uM | -2.460 [-9.73 to 2.72]

4. Secondary Outcome: Long-term Pharmacodynamics (PD) of SC Asfotase Alfa: Pyridoxal-5-phosphate (PLP) Levels
Description: Outcome measure is the change from Baseline in pyridoxal-5-phosphate (PLP) levels. The time period is pre-dose (Baseline from the ENB-002-08 study [NCT00744042]) to the last assessment for each patient in the ENB-003-08 study, which represents up to 90 months of exposure for the combined studies.
Time Frame: Up to 90 Months
Population: Full Analysis Set (All 10 patients enrolled in Study ENB-003-08). Change from Baseline could not be calculated for 2 patients because of non-evaluable samples at Baseline.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 8
ng/mL | -266.200 [-844.30 to 184.00]

5. Secondary Outcome: Effect of SC Asfotase Alfa on Growth: Weight Z-scores
Description: Outcome measure is the change from Baseline in Z-scores for weight. The time period is pre-dose (Baseline from the ENB-002-08 study [NCT00744042]) to the last assessment in the ENB-003-08 study, which represents up to 90 months of exposure in the combined studies.
Time Frame: Up to 90 Months
Population: Full Analysis Set (All 10 patients enrolled in Study ENB-003-08)
Measure: Median (Full Range); unit: Z-score
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 10
Z-score | 2.43 [-2.9 to 5.2]

6. Secondary Outcome: Effect of SC Asfotase Alfa on Growth: Height/Length Z-scores
Description: Outcome measure is the change from Baseline in Z-scores for height/length. The time period is pre-dose (Baseline from the ENB-002-08 study [NCT00744042]) to the last assessment in the ENB-003-08 study, which represents up to 90 months of exposure in the combined studies.
Time Frame: Up to 90 Months
Population: Full Analysis Set (All 10 patients enrolled in Study ENB-003-08)
Measure: Median (Full Range); unit: Z-score
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 10
Z-score | 1.93 [-3.2 to 4.6]

7. Secondary Outcome: Effect of SC Asfotase Alfa on Respiratory Function
Description: Outcome measure is the shift in the proportion of patients requiring respiratory support at their last assessment in Study ENB-003-08 compared with Baseline. The time period is pre-dose (Baseline from the ENB-002-08 study [NCT00744042]) to the last assessment in the ENB-003-08 study, which represents up to 90 months of exposure in the combined studies.
Time Frame: Up to 90 Months
Population: Full Analysis Set (All 10 patients enrolled in Study ENB-003-08)
Measure: Count of Participants; unit: Participants
Groups:
- Asfotase Alfa (Baseline ENB-002-08): Baseline results prior to treatment with asfotase alfa
- Asfotase Alfa (Last Assessment): Results at the last assessment in the ENB-003-08 study.
Arm/Group | Asfotase Alfa (Baseline ENB-002-08) | Asfotase Alfa (Last Assessment)
Number analyzed (Participants) | 11 | 10
Participants
  No respiratory support | 6 | 9
  Supplemental oxygen | 0 | 0
  Continuous positive airway pressure | 1 | 0
  Mechanical ventilation | 3 | 1
  Biphasic positive airway pressure | 0 | 0
  Other | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time the parents/legal guardians signed the ICF for study ENB-003-08 through completion of the patient's participation in the study ENB-003-08.
Arm/Group | Asfotase Alfa
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 9/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asfotase Alfa (N=10)
Cyanosis (Cardiac disorders) | 1 (1)
Congenital bowing of long bones (Congenital, familial and genetic disorders) | 1 (1)
Craniosynostosis (Congenital, familial and genetic disorders) | 4 (5)
Talipes (Congenital, familial and genetic disorders) | 1 (1)
Conductive deafness (Ear and labyrinth disorders) | 1 (1)
Papilloedema (Eye disorders) | 1 (1)
Immediate post-injection reaction (General disorders) | 1 (1)
Medical device complication (General disorders) | 1 (1)
Chronic hepatitis (Hepatobiliary disorders) | 1 (1)
Bacterial tracheitis (Infections and infestations) | 1 (1)
Croup infectious (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (2)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood urea increased (Investigations) | 1 (1)
CSF pressure (Investigations) | 1 (1)
Investigation (Investigations) | 1 (2)
Feeding disorder of infancy or early childhood (Metabolism and nutrition disorders) | 1 (1)
Weight gain poor (Metabolism and nutrition disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (2)
Intracranial pressure increased (Nervous system disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Adenoidal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Central venous catheter removal (Surgical and medical procedures) | 1 (1)
Tracheal fistula repair (Surgical and medical procedures) | 1 (1)
Tracheostomy tube removal (Surgical and medical procedures) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asfotase Alfa (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Microcytosis (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Craniosynostosis (Congenital, familial and genetic disorders) | 2 (5)
Deafness (Ear and labyrinth disorders) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1)
Middle ear disorder (Ear and labyrinth disorders) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Precocious puberty (Endocrine disorders) | 1 (1)
Astigmatism (Eye disorders) | 1 (1)
Conjunctival deposit (Eye disorders) | 1 (2)
Conjunctival hyperaemia (Eye disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 2 (3)
Eye pain (Eye disorders) | 1 (2)
Lacrimation increased (Eye disorders) | 1 (1)
Myopia (Eye disorders) | 1 (1)
Optic disc drusen (Eye disorders) | 1 (1)
Optic nerve disorder (Eye disorders) | 1 (1)
Papilloedema (Eye disorders) | 2 (2)
Visual impairment (Eye disorders) | 2 (4)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (9)
Constipation (Gastrointestinal disorders) | 2 (4)
Dental caries (Gastrointestinal disorders) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 3 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 1 (2)
Gingivitis (Gastrointestinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Teething (Gastrointestinal disorders) | 1 (1)
Tooth loss (Gastrointestinal disorders) | 4 (8)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (14)
Catheter site rash (General disorders) | 1 (1)
Injection site atrophy (General disorders) | 1 (2)
Injection site calcification (General disorders) | 1 (2)
Injection site discolouration (General disorders) | 1 (1)
Injection site erythema (General disorders) | 4 (18)
Injection site haematoma (General disorders) | 2 (2)
Injection site hypertrophy (General disorders) | 2 (8)
Injection site inflammation (General disorders) | 1 (2)
Injection site nodule (General disorders) | 1 (1)
Injection site reaction (General disorders) | 2 (3)
Injection site swelling (General disorders) | 2 (5)
Injection site warmth (General disorders) | 1 (1)
Pain (General disorders) | 3 (4)
Pyrexia (General disorders) | 7 (21)
Vaccination site inflammation (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 2 (2)
Immunisation reaction (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Abscess jaw (Infections and infestations) | 1 (2)
Acute sinusitis (Infections and infestations) | 3 (4)
Bronchitis (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 1 (1)
Croup infectious (Infections and infestations) | 1 (3)
Cystitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (9)
Gastroenteritis viral (Infections and infestations) | 1 (2)
H1N1 influenza (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 3 (7)
Injection site cellulitis (Infections and infestations) | 1 (3)
Laryngitis (Infections and infestations) | 1 (1)
Lice infestation (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2)
Molluscum contagiosum (Infections and infestations) | 1 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Otitis externa (Infections and infestations) | 2 (2)
Otitis media (Infections and infestations) | 6 (23)
Otitis media acute (Infections and infestations) | 1 (1)
Otitis media chronic (Infections and infestations) | 2 (2)
Pharyngitis (Infections and infestations) | 3 (8)
Pneumonia (Infections and infestations) | 5 (7)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Pneumonia primary atypical (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 2 (5)
Sinusitis (Infections and infestations) | 2 (8)
Skin infection (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (6)
Tooth abscess (Infections and infestations) | 2 (2)
Tracheitis (Infections and infestations) | 2 (5)
Upper respiratory tract infection (Infections and infestations) | 8 (77)
Varicella (Infections and infestations) | 2 (2)
Viral infection (Infections and infestations) | 3 (3)
Viral pharyngitis (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (5)
Adverse event following immunisation (Injury, poisoning and procedural complications) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Face injury (Injury, poisoning and procedural complications) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (2)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (2)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood alkaline phosphatase abnormal (Investigations) | 1 (1)
Oxygen saturation decreased (Investigations) | 2 (3)
Staphylococcus test positive (Investigations) | 1 (1)
Urine calcium/creatinine ratio increased (Investigations) | 2 (3)
Vitamin D decreased (Investigations) | 1 (2)
Vitamin D increased (Investigations) | 1 (1)
Abnormal weight gain (Metabolism and nutrition disorders) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemic rickets (Metabolism and nutrition disorders) | 1 (1)
Weight gain poor (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (19)
Scoliosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 5 (14)
Speech disorder developmental (Nervous system disorders) | 2 (2)
Abnormal behaviour (Psychiatric disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anticipatory anxiety (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Fear of needles (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 2 (3)
Nephrocalcinosis (Renal and urinary disorders) | 2 (2)
Renal cyst (Renal and urinary disorders) | 1 (2)
Renal pain (Renal and urinary disorders) | 1 (2)
Breast enlargement (Reproductive system and breast disorders) | 1 (1)
Adenoidal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 (1)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (5)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (3)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria contact (Skin and subcutaneous tissue disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less